CLINICAL TRIAL: NCT03832205
Title: Validation of a Capaciflector Against a Pneumotachometer to Measure Respiratory Rate and a Capaciflector Against Electrocardiography to Measure Heart Rate at Different Anatomical Chest Locations During Cardiopulmonary Exercise Testing
Brief Title: Validation of Respiratory Rate and Heart Rate Measurements by Capaciflectors Placed in Four Locations on the Chest
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CRI0371
Record Dates: First submitted 2018-10-23; First posted 2019-02-06 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Exercise; Respiratory Rate; Heart Rate
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Capaciflector monitoring group: Patients undergoing their pre-planned, routine cardiopulmonary exercise test (CPET). Additional, non-invasive capaciflector monitoring only - no therapeutic intervention.
  Interventions: Device: Capaciflector monitoring

INTERVENTIONS:
Device: Capaciflector monitoring — Non-invasive capaciflector monitoring of respiratory rate and heart rate.

SUMMARY:
In a collaborative project between University Hospital Southampton NHS Trust and the University of Southampton, the investigators have developed a wearable, mobile, non invasive, low-cost, continuous respiratory rate monitor device called a capaciflector.

This study will be the first ever study undertaken to attempt to measure the respiratory rate and heart rate on patients using a capaciflector. Investigators will evaluate whether the correlation between the capaciflector's measurements of respiratory rate and heart rate when compared with the gold standard pneumotachometer and electrocardiogram respectively is high enough to promote its potential future use within a device for clinical practice.

DETAILED DESCRIPTION:
RESEARCH QUESTION/AIM(S)

Will a capaciflector measure the respiratory rate as accurately as a pneumotachometer and the heart rate as accurately as an electrocardiogram?

Objectives:

1. To test the reliability and accuracy of our capaciflector in measuring respiratory rate and heart rate by comparing it with gold standard readings.
2. To assess whether different capaciflector locations around the body are all as accurate as each other.

STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYSIS

Unblinded observational study - for each subject demographic data will be collected: age, gender, height, weight, body mass index.

As well as the routine monitoring devices worn while undergoing a CPET test, the patients will have 4 capaciflectors placed on them as well. These will be placed using hypoallergenic medical grade tape.

* Over the left precordium
* Over the right precordium
* Under the left axilla
* Under the right axilla

Each practical component of the study setup will be delivered consistently by CI Dr Nick Hayward, Student Doctor Alan Doughty, or cardiopulmonary exercise testing (CPET) technicians once the study becomes established. The patient will then undergo a routine CPET and our monitors will not affect what a patient is asked to do as part of the current CPET protocol. If a patient is unable to finish the CPET then their data will still be included.

Raw CPET data will be exported via a feed from the CPET machine and also from the capaciflectors. A laptop computer provided by the University will receive both data feeds. Simultaneous recordings will be taken from each of the capaciflectors at time zero and then at one minute intervals. These anonymous datasets will be stored on the laptop computer. Once the CPET test is completed, the participant's involvement in the study will have ended.

Anonymised raw data analysis comparisons will be made by the Department of Engineering, University of Southampton, in collaboration with the other investigators of this study. There will be no patient identifiable information in any dataset, yet demographic data and raw CPET acquired data will be held securely on the laptop in line with clinical governance requirements of University Hospital Southampton. Statistical support by Dr Helen Moyses of the Clinical Informatics Research Unit, Southampton, will be provided for data analysis at the final stage.

STUDY SETTING

The study will be a single centre study at University Hospital Southampton. Participants will have been recruited from the patients booked for a CPET test prior to them having major surgery. The study will be conducted in the CPET department in the Day Surgery Unit. This is where the CPET for patients routinely takes place.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Able to give informed consent in English
* Able to at least start a CPET test

Exclusion Criteria:

* Absolute contraindications to taking part in CPET:
* Recent (within 5 days) Acute Myocardial Infarction
* Unstable angina
* Uncontrolled arrhythmia causing symptoms or haemodynamic compromise
* Syncope
* Active endocarditis, acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Suspected dissecting or leaking aortic aneurysm
* Uncontrolled asthma
* Arterial desaturation at rest on room air < 85%
* Known allergy to medical grade tape

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing routine clinical cardiopulmonary exercise testing (CPET).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Respiratory rate comparison | Through study completion, an average of one year
  Statistical comparisons between the two methods of measuring respiratory rate
Heart rate comparison | Through study completion, an average of one year
  Statistical comparisons between the two methods of measuring heart rate
Capaciflector location comparison | Through study completion, an average of one year
  Statistical comparisons between the four anatomical chest locations of our capaciflectors

CONTACTS AND LOCATIONS:
Overall Officials: Neil White, PhD, Study Director — University of Southampton
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No personal identifiable data will be shared. Physiological data may be shared with statisticians within the University or University Hospital. Data analysis may be partly conducted by Dr Peter Charlton, Kings College London, UK

REFERENCES:
- [Background] White N. et al. (2017) A Planar Respiration Sensor Based on a Capaciflector Structure. IEEE Sensors Letters vol. 1 no. 4 pp. 1-4 Art no. 6000604. doi: 10.1109/LSENS.2017.2722481. http://ieeexplore.ieee.org/stamp/stamp.jsp?tp=&arnumber=7967772&isnumber=7949374
- [Background] Naranjo-Hernandez D, Talaminos-Barroso A, Reina-Tosina J, Roa LM, Barbarov-Rostan G, Cejudo-Ramos P, Marquez-Martin E, Ortega-Ruiz F. Smart Vest for Respiratory Rate Monitoring of COPD Patients Based on Non-Contact Capacitive Sensing. Sensors (Basel). 2018 Jul 3;18(7):2144. doi: 10.3390/s18072144. PMID 29970861
- [Background] Gerry S, Birks J, Bonnici T, Watkinson PJ, Kirtley S, Collins GS. Early warning scores for detecting deterioration in adult hospital patients: a systematic review protocol. BMJ Open. 2017 Dec 3;7(12):e019268. doi: 10.1136/bmjopen-2017-019268. PMID 29203508
- [Background] Effects of current on human beings and livestock - Part 1: General Aspects, section 4.5.4 (1993) Bureau of Indian Standards, New Delhi. http://questin.org/sites/default/files/standards/is.8437.1.1992_0.pdf
- [Derived] Hayward N, Shaban M, Badger J, Jones I, Wei Y, Spencer D, Isichei S, Knight M, Otto J, Rayat G, Levett D, Grocott M, Akerman H, White N. A capaciflector provides continuous and accurate respiratory rate monitoring for patients at rest and during exercise. J Clin Monit Comput. 2022 Oct;36(5):1535-1546. doi: 10.1007/s10877-021-00798-7. Epub 2022 Jan 18. PMID 35040037